CLINICAL TRIAL: NCT06377423
Title: Randomized Clinical Trial on Direct Composite and Indirect Ceramic Laminate Veneers in Multiple Diastema Closure Cases: 2-years Follow-up
Brief Title: Comparison Between Direct Composite and Indirect Ceramic Laminate Veneers in Multiple Diastema Closure Cases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prince Sattam Bin Abdulaziz University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A54678775
Record Dates: First submitted 2024-04-11; First posted 2024-04-22 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Dental Leakage
Keywords: Ceramics; Composite; Randomized clinical trial; diastema closure
MeSH Terms: conditions — Dental Leakage | interventions — Fluorescent Antibody Technique, Direct

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Estelite esteria composite (Experimental): Half of the patients received composite veneers using direct method
  Interventions: Procedure: Direct technique
- IPS Emax press ceramic (Experimental): Half of the patients received ceramic veneers using indirect technique
  Interventions: Procedure: Indirect technique

INTERVENTIONS:
Procedure: Direct technique — The composite was placed directly using free-hand technique
  Arms: Estelite esteria composite
Procedure: Indirect technique — The ceramic was placed using indirect method via laboratory casts
  Arms: IPS Emax press ceramic

SUMMARY:
Thus, the present study aimed to evaluate the longevity of direct composite compared to indirect ceramic laminate veneers in multiple diastema closure cases using USPHS criteria. The formulated null hypothesis was that there is no significant difference in the clinical performance of direct composite and indirect ceramic laminate veneers in multiple diastema closure cases over two years.

DETAILED DESCRIPTION:
Restorative materials and curing device In the current study, the manufacturer's instructions were followed for the use of the nanofilled composite resin (Estelite Asteria, Tokuyama Dental, Japan) for direct laminate veneers and IPS e.max Press (Ivoclar Vivadent, Amherst, NY, USA) for indirect laminate ceramic veneers. A light curing device with an output density of 655 mW/cm2 (LED Bluephase C5, Ivoclar, Vivadent, Amherst, NY, USA) was used. Demetron LED light meters were used to measure the light curing unit's intensity regularly (Demetron Research Corp., Danbury, CT, USA). Brand name, description, chemical composition, and manufacturers of the materials are presented in Table 1.

Study design, blinding & randomization The Consolidated Standards of Reporting Trials statement was adhered to in the description of the experimental design. This study was a randomized controlled clinical trial that was double-blinded for both trial participants and outcome assessors. Randomization was performed using the flip of a coin for the choice of material. Using computerized sequence generating (www. randomizer.org), participants were divided into two groups with a 1:1 allocation ratio.

ELIGIBILITY:
Inclusion Criteria:

* Patients needed diastema closure.
* Patients with normal and full occlusion.
* Patients must have a good oral hygiene.
* Patients with a tooth respond positively to an electric pulp tester.

Exclusion Criteria:

* High caries risk patients with extremely poor oral hygiene.
* Patients with periodontally-involved teeth.
* Patients with heavy bruxism habits and clenching.
* Patients involved in orthodontic treatment.

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-01-10 (Actual)

PRIMARY OUTCOMES:
Percentage % of patients with marginal staining | 2 years after restoration procedure
  The percentage of marginal staining in patients was clinically assessed using USPHS criteria. Restorations were given scores from 0 to 5

CONTACTS AND LOCATIONS:
Overall Officials: Abdallah Elshehri, Phd, Study Director — Dept. of Conservative Dental Sciences, College of Dentistry, Prince Sattam Bin Abdulaziz University
Locations (1):
- Ali Elkaffas, Al Kharj, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes
Plan can be shared with other researchers
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available within 6 months for 5 years
Access Criteria: For anyone